CLINICAL TRIAL: NCT04579887
Title: Unravelling Dysfunctional Brain Networks in Patients With Parkinson's Disease Suffering From Presence Hallucination
Brief Title: Presence Hallucination in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olaf Blanke (Other)
Collaborators: University Hospital, Geneva (Other); Centre Hospitalier Universitaire Vaudois (Other); Insel Gruppe AG, University Hospital Bern (Other); Hôpital du Valais (Other)
Responsible Party: Sponsor-Investigator, Olaf Blanke, Professor Doctor, Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PD_PH
Record Dates: First submitted 2020-07-15; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease Psychosis
Keywords: Parkinson; fMRI; connectivity; hallucinations; psychosis; presence hallucination
MeSH Terms: conditions — Hallucinations; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain changes triggered by PH induction in Parkinson's disease (Experimental): Clinical and neuropsychological evaluations + Sensorimotor task for PH-induction
  Interventions: Other: Brain changes triggered by PH induction in Parkinson's disease patients with presence hallucinations

INTERVENTIONS:
Other: Brain changes triggered by PH induction in Parkinson's disease patients with presence hallucinations — Parkinsonian patients will undergo a two distinct experimental sessions, conducted in two separate days. In day 1, they will complete a series of validated and lab-tailored clinical evaluations, alongside with semi-structured interviews. These tests are designed to assess, the extent of the movement disorder, the predominance of positive symptoms and presence hallucination, potential cognitive impairment, amongst other relevant measures, for sleep assessment, loneliness, apathy and depression. In day 2 patients will perform the described robotic manipulation task in the MRI.

SUMMARY:
Investigation on how robotically mediated sensorimotor stimulation induces and triggers presence hallucinations in patients with Parkinson disease

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is primarily known and characterized by motor symptoms such as tremor, rigidity and bradykinesia. However, a significant number of non-motor symptoms also accompany the unfolding of this disease. In fact, hallucinations are experienced by approximately 60% of the patients. The most common and amongst one of the earliest hallucinations in Parkinson's Disease, is the Presence Hallucination (PH), i.e., the strange sensation of perceiving someone behind when no one is actually there. In the present study the researchers aim at investigating the behavioural and neural mechanisms underlying symptomatic PH in PD. To do so the researchers intend to induce the PH in a repeated and controlled manner in the MRI scanner, with an extensively verified paradigm which gives rise to this sensation by means of robotically-mediated sensorimotor stimulation. This setup has in fact been shown to trigger the occurrence of symptomatic PH in these patients. The possibility to induce PH while the patient is in the MRI will allow the researchers to investigate online the brain networks associated with it.

With analysis on the fine brain connectivity changes during PH-induction, the investigators intend to pinpoint the exact mechanism behind the appearance of this hallucination in these patients, in a similar fashion to previous work with the PH-induction in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease
* Able to understand instructions and provide informed consent.
* Native speaking language of experimental site (or acquisition of language of experimental site before 6 years old).
* Montreal Cognitive Assessment (Nasreddine & Patel, 2016) with score ≥ 22.
* Able to manipulate the robotic device.

Exclusion Criteria:

* Neurological comorbidities other than Parkinson's disease (e.g. Alzheimer's disease, vascular dementia, multiple sclerosis, stroke, traumatic brain injury, epilepsy, chronic migraine, etc.)
* History or current condition of substance abuse and/or dependence (e.g., alcohol, drugs).
* Suffering from or diagnosed with psychiatric illnesses according to DSM-V criteria (e.g., schizophrenia, bipolar disorders, autism, personality disorders, phobia etc.).
* Family history (1st and 2nd degree) of psychiatric disorders (e.g., schizophrenia or bipolar disorders).
* Severe somatic illnesses (e.g., cancer).
* Severe tremors or physical disability preventing optimal use of robotic device.
* Participating in a pharmacological study.
* Local or general anaesthesia 30 days prior experiment
* Inability to provide informed consent (legal guardianship)
* The following are due to the MRI scanner: body weight exceeding 160kg, implanted metallic devices, foreign metallic objects, unstable angina, cardio-vascular diseases, tattoos with metallic components, external metallic objects, claustrophobia, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
fMRI bold signal response during robotic manipulation | Approximately 45 minutes during each participant's experimental session in arm 1
  Analysis of changes of BOLD activity during the asynchronous condition as compared to the synchronous condition
Sensitivity to the induction bodily illusions of Presence Hallucination, Passivity experiences, loss of agency, and control questions, through lab-tailored questionnaires (7-point Likert-scale) | Approximately 5 minutes at the end of each participant's experimental session in arm 1
  Note that for the assessment of the sensitivity of each patient to the induction of the presence hallucination, passivity sensations, loss of agency, and control questions, the patients will perform two manipulations with the robotic system described in the introduction, in both the synchronous and asynchronous conditions

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Blanke, Principal Investigator — Ecole Polytechnique Fédérale de Lausanne
Locations (4):
- Switzerland (4):
  - Inselspital, Bern
  - Campus Biotech, Geneva
  - HUG, Geneva
  - Hôpital du Valais, Sion

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalia LV, Lang AE. Parkinson's disease. Lancet. 2015 Aug 29;386(9996):896-912. doi: 10.1016/S0140-6736(14)61393-3. Epub 2015 Apr 19. PMID 25904081
- [Background] Postuma RB, Berg D. Advances in markers of prodromal Parkinson disease. Nat Rev Neurol. 2016 Oct 27;12(11):622-634. doi: 10.1038/nrneurol.2016.152. PMID 27786242
- [Background] Wood RA, Hopkins SA, Moodley KK, Chan D. Fifty Percent Prevalence of Extracampine Hallucinations in Parkinson's Disease Patients. Front Neurol. 2015 Dec 21;6:263. doi: 10.3389/fneur.2015.00263. eCollection 2015. PMID 26733937
- [Background] Diederich NJ, Fenelon G, Stebbins G, Goetz CG. Hallucinations in Parkinson disease. Nat Rev Neurol. 2009 Jun;5(6):331-42. doi: 10.1038/nrneurol.2009.62. PMID 19498436
- [Background] Fenelon G, Soulas T, Cleret de Langavant L, Trinkler I, Bachoud-Levi AC. Feeling of presence in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2011 Nov;82(11):1219-24. doi: 10.1136/jnnp.2010.234799. Epub 2011 May 7. PMID 21551471
- [Background] Blanke O, Pozeg P, Hara M, Heydrich L, Serino A, Yamamoto A, Higuchi T, Salomon R, Seeck M, Landis T, Arzy S, Herbelin B, Bleuler H, Rognini G. Neurological and robot-controlled induction of an apparition. Curr Biol. 2014 Nov 17;24(22):2681-6. doi: 10.1016/j.cub.2014.09.049. Epub 2014 Nov 6. PMID 25447995
- See also: Bernasconi F, Blondiaux E, Potheegadoo J, Stripeikyte G, ..., Blanke O (2020) sensorimotor hallucinations in Parkinson's disease — https://www.biorxiv.org/content/10.1101/2020.05.11.054619v1